CLINICAL TRIAL: NCT03477799
Title: The Effect of Transcranial Direct Current Stimulation on Decision Making and Cognitive Flexibility in Gambling Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ahmet Zihni Soyata, Resident, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 71146310-511.06-E368557
Record Dates: First submitted 2018-03-13; First posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Gambling Disorder
Keywords: gambling disorder; cognition
MeSH Terms: conditions — Gambling | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator): anodal stimulation over the right dlPFC
  Interventions: Device: Transcranial direct current stimulation
- Sham (Placebo Comparator): sham stimulation over the right dlPFC
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Transcranial direct current stimulation (tDCS) is a safe method for non-invasively modulating cortical excitability through the use of weak electrical currents (usually of 1-2 mA) circulating between two scalp electrodes (i.e., an anode and a cathode) placed over the target cortical regions. The effects of tDCS on brain activity are polarity-dependent, such that anodal stimulation generally enhances cortical excitability by depolarizing cell membranes and increasing neuronal firing rates, while cathodal stimulation generally results in the opposite effect. Because of its neural effects, tDCS has been increasingly used to gauge the functional relationship between cognitive/behavioural dimensions and putatively relevant neurocircuitry

SUMMARY:
The investigators conducted a double-blind randomised sham-controlled study. Upon enrollment into the study, participants were randomly assigned to one of two conditions: (i) active group: anodal stimulation over the right dlPFC (n = 10) or (ii) sham stimulation group (n = 10). Participants and raters were blinded to the condition.

Subsequently, the participants were administered the IGT and the Wisconsin Card Sorting Test by a trained neuropsychologist in a quiet laboratory. A computerized version of standard IGT was used. The order of the tasks performed in a single session was randomised.

After the psychiatric and neurocognitive assessment, participants received three sessions of 20-minute active or sham anodal tDCS (once a day, every other day).

Wisconsin Card Sorting Test and a modified version of Iowa Gambling Test were readministered after the last application. The order of the tasks was randomized again. A brief questionnaire on study blinding was also administered. Safety was assessed through open-ended questions based on the tDCS adverse events questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Participants meeting Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for gambling disorder
* Being right-handed
* Being 18-65 years old
* Being drug-free

Exclusion Criteria:

* Current DSM-5 diagnosis of major depressive disorder
* Current or previous DSM-5 diagnosis of alcohol and substance use disorders, schizophrenia, bipolar disorder, or other psychotic disorder
* Drug Use in the past 4 weeks of any medication with known pro-convulsant action or current regular use of any psychotropic medications (benzodiazepines, antipsychotic medications, tricyclic antidepressants, anti-epileptics, mood stabilizers)
* Any history of any clinically significant neurological disorder, including organic brain disease, epilepsy, stroke, brain lesions, multiple sclerosis, previous neurosurgery, or personal history of head trauma that resulted in loss of consciousness for > 5 minutes and retrograde amnesia for > 30 minutes,
* The presence of mental retardation diagnosis (previously identified)
* Any personal or family history (1st degree relatives) of seizures other than febrile childhood seizures
* Illiteracy, deficient language or refusal to participate.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Changes in the Iowa Gambling Task net score | Baseline, after tDCS treatment
  Iowa Gambling Task net score is the total score of the task (between -100 and 100) that generally assesses the decision making under ambiguity, but also assesses the decision making under risk at the later stages. Higher scores in the task represents better decision making and healthy people generally have scores above 8-10 in the task.
Changes in the number of perseverative errors in Wisconsin Card Sorting Task | Baseline, after tDCS treatment
  Wisconsin Card Sorting Task is the widely used task to assess frontal lobe functions such as cognitive flexibility, set shifting and abstraction abilities. The participants were required to match response cards to 4 stimulus cards along 1 of 3 dimensions (colour, form or number) on the basis of verbal feedback (correct or incorrect). The participants were not given any information about the dimensions. After sorting a series of 10 cards in 1 category, participants were asked to sort the cards in a different category. The number of perseverative errors in Wisconsin Card Sorting Task is the most robust variable of the task to assess cognitive flexibility. Higher scores show an impairment of cognitive flexibility

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Z Soyata, Principal Investigator — Resident
Locations (1):
- Ahmet Zihni Soyata, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Soyata AZ, Aksu S, Woods AJ, Iscen P, Sacar KT, Karamursel S. Effect of transcranial direct current stimulation on decision making and cognitive flexibility in gambling disorder. Eur Arch Psychiatry Clin Neurosci. 2019 Apr;269(3):275-284. doi: 10.1007/s00406-018-0948-5. Epub 2018 Oct 26. PMID 30367243